CLINICAL TRIAL: NCT02136615
Title: Does Hyperbaric Oxygen Therapy Lead to a Sustained Increase in Insulin
Brief Title: Does Hyperbaric Oxygen Therapy Lead to a Sustained Increase in Insulin Sensitivity?
Acronym: HOTAIR3
Status: Completed | Type: Observational
Sponsor: University of Adelaide (Other)
Collaborators: Australasian Hyperbaric & Diving Medicine Research Trust (Unknown)
Responsible Party: Principal Investigator, A/Prof Leonie Heilbronn, ARC Future Fellow, University of Adelaide
Other Study IDs: HREC/14/RAH/118
Record Dates: First submitted 2014-05-02; First posted 2014-05-13 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Overweight and Obesity; Insulin Sensitivity
Keywords: hyperbaric oxygenation; insulin sensitivity; human; inflammation; adipose tissue
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, adipose tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- overweight and obese male volunteers: BMI between 23-40 kg/m2

SUMMARY:
In a recent series of studies performed by our group, we have shown that exposure to hyperbaric oxygen (HBOT) leads to an increase in insulin sensitivity in male subjects and that this improvement can be measured in all men, not just those with diabetes. The aim of this study is to investigate the time course of this effect and explore the mechanisms involved when exposure to HBOT induces an increase in peripheral insulin sensitivity.

Aims:

1. To determine whether the insulin sensitising effect of HBOT is apparent 24-hours after an HBO session.
2. To examine mechanisms underpinning the increase in insulin sensitivity following HBOT.

DETAILED DESCRIPTION:
All participants will attend the Hyperbaric Medicine Unit on 5 occasions. Day 1 will be for baseline assessment. Days 2 to 5 will be on consecutive days the following week. An overnight fast will be required prior to each day.

Day 1. Baseline assessment. The participant will attend after an overnight fast at 0830 for frequently sampled intravenous glucose tolerance test (FSIGT). Two IV lines will be placed and baseline blood samples (30ml) are drawn for measurement of gluco-regulatory hormones and metabolites at time 0. A glucose bolus is then administered through the antecubital vein IV (300mg/kg, 25% Dextrose infused over 1-minute) at time 0. Blood sampling (3ml) is then performed at 2,4,6,8,10,12,14,16,19,22,25,30,40,50,60,70,90,120,150,180 minutes after the completion of the glucose bolus. Each blood sample is analysed for glucose and insulin. Total blood collected during this procedure is approximately 60mls. A urine sample will be collected. A meal will be provided.

Day 2. The following week, the participant will attend at 0800 after an overnight fast. They will then be placed supine on a bed and a subcutaneous adipose tissue biopsy will be performed using the technique of Bergstrom: after cleansing the skin on the abdomen lateral to the umbilicus with chlorhexidine solution, and placing a fenestrated drape, anaesthesia is administered (5mL of Xylocaine 2%, no adrenaline). A 7.5mm incision is made in the skin (#11 scalpel) and a 5mm Bergstrom needle inserted to collect approximately 250mg of adipose tissue with suction. Two or three passes will be used to obtain approximately 500mg of adipose tissue. The sample is washed in sterile phosphate buffer solution and snap frozen in liquid nitrogen. Upon completion of the biopsy the incision is closed with a sterile bandage, a sterile dressing applied and pressure is applied for 10-minutes. Blood will be taken for glucose, insulin and inflammatory markers (30mls). The participant will then sit in a chair for 2-hours during a routine HBOT session from 0830-1030 (10:90:30 profile). After the first HBOT, a further blood sample will be taken for inflammatory markers. Food will be provided.

Day 3. After an overnight fast, the participant will undergo a second routine HBOT session from 0830-1030, followed by a second fat tissue biopsy. Blood will be taken for glucose, insulin and inflammatory markers (30mls) before and after the HBOT. Food will be provided.

Day 4. After an overnight fast, the participant will undergo a third HBOT session from 0830-1030. This will be undertaken simultaneously with a FSIGT. The IV glucose bolus will be administered at the beginning of the HBOT once the hyperbaric chamber has reached treatment pressure (2 atmospheres absolute). On completion of the FSIGT, a meal will be provided.

Day 5. After an overnight fast, the participant will attend at 0830 for a fourth blood sample for inflammatory markers. An FSIGT will be performed in room air outside the hyperbaric chamber. A meal will be provided. A urine sample will be collected.

With blood taken during three FSIGTs together with 5 blood samples taken for inflammatory markers, a total of about 330 mls of blood will be drawn over 9 days.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 (no specific upper age limit)
* All participants will be assessed by a hyperbaric physician to determine fitness to enter the hyperbaric chamber - the standard clinical criteria of the Hyperbaric Medicine Unit will be used

Exclusion Criteria:

* Personal history of Diabetes or major psychiatric disorders,
* use of prescribed or non-prescribed medications which may affect glucose homeostasis (eg steroids)
* uncontrolled asthma, current fever, upper respiratory infections
* individuals who regularly perform high intensity exercise (>2 week)
* current intake of > 140g alcohol/week
* current smokers of cigarettes/cigars/marijuana
* current intake of any illicit substance
* experience claustrophobia in confined spaces
* has donated blood within past 3-months
* has been involved in any other study within the past 3-months
* unable to comprehend study protocol
* any other contraindication to HBOT (eg Eustachian tube dysfunction making middle ear inflation ineffective)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity as measured by FSIGT | Baseline, Day 5
  24-hours after the last HBOT

SECONDARY OUTCOMES:
Changes in inflammatory markers from blood | Baseline, Day 2
  After first HBOT
Change in insulin sensitivity by FSIGT | Baseline, Day 4
  During third and final HBOT
Changes in inflammatory markers from blood | Baseline, Day 3
  After second HBOT
Changes in inflammatory markers from blood | Baseline, Day 5
  24-hours after final HBOT

OTHER OUTCOMES:
Changes in gene expression from adipose tissue | Baseline, Day 3
  After two HBOT

CONTACTS AND LOCATIONS:
Overall Officials: Leonie K Heilbronn, PhD, Principal Investigator — University of Adelaide, Discipline of Medicine
Locations (1):
- Hyperbaric Medicine Unit, Royal Adelaide Hospital, Adelaide, South Australia, Australia

REFERENCES:
- [Background] Wilkinson D, Chapman IM, Heilbronn LK. Hyperbaric oxygen therapy improves peripheral insulin sensitivity in humans. Diabet Med. 2012 Aug;29(8):986-9. doi: 10.1111/j.1464-5491.2012.03587.x. PMID 22269009